CLINICAL TRIAL: NCT02926326
Title: An Open-label, Single-sequence Study to Evaluate the Effect of Azithromycin on BCT197 Exposure in Healthy Male Subjects
Brief Title: The Effect of Azithromycin on BCT197 Exposure in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mereo BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBCT102
Record Dates: First submitted 2016-09-28; First posted 2016-10-06 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Interaction
Keywords: Healthy Male volunteers
MeSH Terms: interventions — acumapimod; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Period 1 and Period 2 (Other): Period 1 - BCT197 14mg on Day 1
  Period 2 - BCT 197 14mg on Day 1 and Azithromycin 500mg on Day 1,2 and 3
  Interventions: Drug: BCT197; Drug: Azithromycin

INTERVENTIONS:
Drug: BCT197 — A single dose of BCT197
  Other Names: Acumapimod
Drug: Azithromycin — 3 daily doses of Azithromycin

SUMMARY:
An open-label, single-sequence study to evaluate the effect of azithromycin on BCT197 exposure in healthy male subjects.

DETAILED DESCRIPTION:
This will be an open study conducted in healthy male subjects at a single centre. Each subject will participate in a screening visit and 2 study periods. At the first study period, all subjects will receive a single dose of BCT197 and at study period 2, all subjects will receive 3 daily doses of azithromycin and a single dose of BCT197.

ELIGIBILITY:
Inclusion Criteria

* Healthy male subjects.
* Non-smokers (including e-cigarettes).
* Body mass index (BMI) ≥ 18 and ≤ 30 kg/m2.
* Willing to use highly effective barrier contraception methods.
* Male subjects must not donate sperm during the study.

Exclusion Criteria

* Any subjects with pre-existing active skin disease.
* Laboratory values at screening which are deemed to be clinically significant.
* Volunteers with abnormal liver function tests.
* 12 Lead ECG with QTcF >450 msec.
* Allergy to any of BCT197 excipients.
* Known hypersensitivity or intolerance to azithromycin.
* Taking medications known to cause QTc prolongation.
* Positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
* Any clinically significant illness within 30 days prior to study drug administration.
* Volunteers who, in the opinion of the Investigator, are unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Maximum Measurable Plasma Concentration (Cmax) BCT197 in the presence and absence of Azithromycin. | Pre-dose to Day 15
  Period 1: Pre-dose and 1, 2, 4, 6, 12, 24, 36, 48, 72,96, 144, 168 hours post BCT197 dose on Day 1.
  Period 2: Pre BCT197 dose, 1, 2, 4, 6, 12, 24, 36, 48,72, 96,144, 168 and 336 hours post BCT197 dose on Day 1.
Area under the plasma concentration-time curve (AUC) BCT197 in the presence and absence of Azithromycin. | Pre-dose to Day 15
  Period 1: Pre-dose and 1, 2, 4, 6, 12, 24, 36, 48, 72,96, 144, 168 hours post BCT197 dose on Day 1.
  Period 2: Pre BCT197 dose, 1, 2, 4, 6, 12, 24, 36, 48,72, 96,144, 168 and 336 hours post BCT197 dose on Day 1.

SECONDARY OUTCOMES:
The number of adverse events during administration of BCT197 alone and in the presence of Azithromycin. | Day 1 to Day 22

OTHER OUTCOMES:
Corrected QT interval of the electrocardiogram (QTc). | Pre-dose to Day 15
  Period 1: Pre-dose, 1, 2, 4, 6, 8, 24 and 168 hours post BCT197 dose on Day 1.
  Period 2: -22 hours, -16 hours, pre-dose azithromycin, 2, 4, 6, 8, 24, 168 and 336 hours post-dose (BCT197 on Day 1).

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Parkin, PhD FRCP, Study Director — Mereo BioPharma
Locations (1):
- BioKinetic Europe Ltd, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No